CLINICAL TRIAL: NCT04366336
Title: Blood Flow Restriction Training Vs Standard Physical Therapy Following Total Knee Arthroplasty Prospective Intervention Study (Blood Flow Restriction Training: BFRT)
Brief Title: BFRT vs Standard PT After Total Knee Arthroplasty
Acronym: BFRT-TKA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Several SubInvestigators have left Institution
Sponsor: Norton Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-N0153
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Blood Flow Restriction Training; Quadriceps Strengthening
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Flow Restriction Training (Experimental): Blood flow restriction training (BFRT) uses a specialized tourniquet system to restrict arterial inflow and venous outflow to the limb during low-load resistance exercise.
  BFRT involves placing the pressure cuff before the start of therapeutic exercises.
  Therapeutic exercise, including but not limited to: movement re-education, balance, and functional strength training; Manual Physical Therapy including but not limited to passive range of motion (therapist will move your knee without your help), joint mobilization, soft-tissue mobilization and static stretching
  Interventions: Procedure: Blood Flow Restriction Training
- Standard Physical Therapy (Active Comparator): Subjects will receive American College of Sports Medicine guided-strength training Therapeutic exercise, including but not limited to: movement re-education, balance, and functional strength training; and Manual Physical Therapy including but not limited to passive range of motion (therapist will move your knee without your help), joint mobilization, soft-tissue mobilization and static stretching
  Interventions: Procedure: Standard Physical Therapy

INTERVENTIONS:
Procedure: Blood Flow Restriction Training — Same as Standard PT with the exception that BFRT involves placing the pressure cuff before the start of therapeutic exercises
  Arms: Blood Flow Restriction Training
Procedure: Standard Physical Therapy — Therapeutic exercise, including but not limited to: movement re-education, balance, and functional strength training; and Manual Physical Therapy including but not limited to passive range of motion (therapist will move your knee without your help), joint mobilization, soft-tissue mobilization and static stretching
  Arms: Standard Physical Therapy

SUMMARY:
Background Blood flow restriction training (BFRT) uses a specialized tourniquet system to restrict arterial inflow and venous outflow to the limb during low-load resistance exercise. BFRT has the potential to augment strength gains for rehabilitation patients who are unable to tolerate high intensity resistance training.

Objective To determine if BFRT will accelerate the recovery of thigh muscle function and strength in post-operative TKA compared to a standard post-operative rehabilitation protocol.

Primary Outcome Measures:

Quadriceps Strength: dynamometry (hand held)

Secondary Outcomes Measures:

Patient Reported Outcomes Knee Injury and Osteoarthritis Outcome Score, Jr Veterans Rand -12 Functional Measures Timed stair ascent Four square Test 5x Sit to Stand Test

Study Design Open label randomized clinical trial with a 1:1 allocation in random sized blocks

Sample Size Based on a Pre-TKA Quadriceps Maximal Voluntary Isometric Contraction mean of 18 with a standard deviation of 8, expecting a 20% improvement of MVIC with BFRT compared to standard Physical Therapy, with an α of 0.05 and β of 0.20 (80% power), the sample size is 63 in each arm. To account for a 20% drop-out rate, a total of 75 subjects will be enrolled in each arm Study Arms Control arm: Subjects will receive American College of Sports Medicine guided-strength training Experimental: Subjects will receive BFRT strength training as part of their post-operative physical therapy program for two months during normal post-op rehab.

DETAILED DESCRIPTION:
Background Blood flow restriction training (BFRT) uses a specialized tourniquet system to restrict arterial inflow and venous outflow to the limb during low-load resistance exercise. BFRT has the potential to augment strength gains for rehabilitation patients who are unable to tolerate high intensity resistance training.

Objective To determine if BFRT will accelerate the recovery of thigh muscle function and strength in post-operative TKA compared to a standard post-operative rehabilitation protocol.

Primary Outcome Measures:

Quadriceps Strength: dynamometry (hand held)

Secondary Outcomes Measures:

Patient Reported Outcomes Knee Injury and Osteoarthritis Outcome Score, Jr Veterans Rand -12 Functional Measures Timed stair ascent Four square Test 5x Sit to Stand Test

Study Design Open label randomized clinical trial with a 1:1 allocation in random sized blocks

Sample Size Based on a Pre-TKA Quadriceps Maximal Voluntary Isometric Contraction mean of 18 with a standard deviation of 8, expecting a 20% improvement of MVIC with BFRT compared to standard Physical Therapy, with an α of 0.05 and β of 0.20 (80% power), the sample size is 63 in each arm. To account for a 20% drop-out rate, a total of 75 subjects will be enrolled in each arm

Study Arms Control arm: Subjects will receive American College of Sports Medicine guided-strength training Experimental: Subjects will receive BFRT strength training as part of their post-operative physical therapy program for two months during normal post-op rehab.

ELIGIBILITY:
Inclusion Criteria:

* Status post primary TKA and cleared by surgeon for Physical Therapy.
* Ages 50-79 years old
* Able to participate fully in PT
* Primary cruciate retaining or posterior stabilized TKA.
* Knee Range of Motion of surgical extremity is a minimum of 5° on full extension to 90° on full flexion

  • Exclusion Criteria:
* Unable to consent for study participation
* Unable to participate in preoperative testing
* Any ligamentous or osseous reconstruction at time of surgery that limits weight bearing
* History of Deep Vein Thrombosis
* Injury or recent procedure to uninvolved extremity within 6 months
* History of endothelial dysfunction
* History of Peripheral Vascular Disease including varicose veins
* Easy bruisability
* TKA is revision
* History of surgical wound complication on involved extremity
* History of stroke
* History of dementia
* History of neuromuscular disorder
* History of Chronic Obstructive Pulmonary Disease
* History of diabetes mellitus with neuropathy
* History of previous intra-articular fracture of involved extremity causing surgical fixation
* History of sickle cell trait/disease
* Previous participation in BFRT
* Any surgical procedure affecting their ability to complete all PT sessions or testing.
* History of functionally limiting arthritis in non-surgical Lower Extremity
* Prior contralateral Total Knee Arthroplasty
* Prior Total Hip Arthroplasty
* Positive pregnancy test
* Enrollment into another clinical research trial

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Quadriceps Strength | 12 weeks post-op
  Quadriceps Strength measured using a handheld dynamoneter

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score, Jr, | Pre-Op, 6 and 12 weeks and 12 months post-op
  Knee Injury and Osteoarthritis Outcome Score, Jr,
Veterans Rand -12 | Pre-Op, 6 and 12 weeks and 12 months post-op
  Veterans Rand -12
Four square Test | Pre-Op, 6 and 12 weeks post-op
  Subject will be asked to walk forward, sideways, backward and sideways over four squares.
5x Sit to Stand Test | Pre-Op, 6 and 12 weeks and 12 months post-op
  Subject will be asked to sit in a chair with back straight and feet on a flat surface positioned about shoulder width apart, arms crossed at chest and asked to stand up and sit down five times.
Quadriceps Strength | 6 weeks post-op
  Quadriceps Strength measured using a handheld dynamoneter
Quadriceps Strength | 12 months post-op
  Quadriceps Strength measured using a handheld dynamoneter

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Stimac, MD, Principal Investigator — Norton Healthcare
Locations (1):
- Norton Healthcare, Louisville, Kentucky, United States